CLINICAL TRIAL: NCT05981872
Title: EFFECT OF COGNITIVE BEHAVIORAL THERAPY ON DEPRESSION AND QUALITY OF LIFE IN PATIENTS WITH POST COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Allaa Ashraf Maher Mohammed Elfwey, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Rehacom on post covid
Record Dates: First submitted 2023-08-05; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Post-COVID-19 Syndrome
Keywords: Rehacom; post covid-19; cognitive rehabilitation; depression; Quality of life
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Study group (A) which will include 18 patients who will receive cognitive rehabilitation (Rehacom ) and selected physical therapy program.
  Control group (B) which will include 18 patients who will receive only selected physical therapy program
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- post covid-19 patients with neurological symptoms as study group (Experimental): •Study group (A) will receive cognitive rehabilitation (Rehacom ) for 30 minutes and selected physical therapy program(that included aerobic, strength, and balance training for 30 minutes, with total duration 60 minutes. 3 sessions per week for 12 weeks.
  Interventions: Behavioral: rehacom
- post covid-19 patients with neurological symptoms as control group (Active Comparator): Control group (B) which will include 18 patients who will receive only selected physical therapy program (that included aerobic, strength, and balance training ).
  The treatment will conducted for 60 minutes, 3 sessions per week for 12 weeks
  Interventions: Behavioral: rehacom

INTERVENTIONS:
Behavioral: rehacom — Rehacom was carried out at the cognition laboratory at Faculty of physical therapy, Cairo University for training of figural memory, attention concentration.
  1. Attention concentration training consists of 24 levels of difficulties .
  2. Figural memory training consists of 9 levels of difficulties. In the training session, every patient was starting training from level one and when the patient successfully finished the level, the training then Progress to the level of difficulty.
  Other Names: cognitive behavioral therapy

SUMMARY:
The goal of this clinical trial is to test the effect of Rehacom on depression and Quality of life in post covid -19 patients. The main question it aims to answer is:

• Is a cognitive rehabilitation therapy will improve depression and quality of life in patients with post COVID-19? Researchers will compare Rehacom with exercise therapy to see if rehacom can improve depression and quality of life in patients with post COVID-19 neuropsychological problems.

DETAILED DESCRIPTION:
Purpose of the study:

* To investigate the effect of cognitive rehabilitation therapy on depression in post COVID-19 patients.
* To investigate the effect of cognitive rehabilitation therapy on quality of life in post COVID-19 patients.

Significance of the study:

•There is growing evidence that individuals with COVID-19 disease can develop a range of neurological complications including cognitive and neuropsychiatric symptoms . Cognitive rehabilitation essential in improving quality of life with Introduction of new neuropsychological rehabilitation tools based on the latest developments in computer sciences.

This study aims to investigate the RehaCom as a cognitive rehabilitation program on depression and quality of life in patients suffer from post COVID-19 neuropsychological problems.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be selected according to following criteria:

  1. Patients from both genders (male and female).
  2. The age of participants ranged from 30 to 45 years .
  3. The patients had score more than 24 according to Mini mental state examination (MMSE).
  4. Patient muscle power not less than grade 3 .
  5. Patients are ambulant.
  6. Patients with confirmation of previous covid19 infection PCR TEST.
  7. Participants were required to live in Egypt during the pre-covid and COVID-19 pandemic.
  8. Patients meeting the guide line of world health organization (WHO) of long/post-covid 19 syndromes.
  9. Patients are "long-haulers" those who history of probable or confirmed SARS-CoV-2 infection; usually within three months from the onset of COVID-19, and last more than two months

Exclusion Criteria:

* The patients will be excluded if they have any of the following:

  1. Patient previously diagnosed with depression and currently taking medication.
  2. patient had prior cognitive impairment.
  3. Illiterate patients.
  4. patient had experienced another major stressful event (e.g., divorce, bereavement) in the past year.
  5. Checking comorbidities (sum of hypertension, diabetes, arrhythmia, myocardial infarction, Chronic Obstructive Pulmonary Disease/Asthma.
  6. Mild cognitive impairment, dementia, other neurodegenerative diseases, stroke, depression,
  7. Osteoarthritis , low back pain and prevalence of polypharmacy (5 or more drugs) at admission.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
The Mini- Mental State Examination (MMSE) | The MMSE is easily administered and requires only 5-10 minutes to complete depending on the impairment of the individual
  The Mini- Mental State Examination (MMSE) was designed to provide a standardized, brief and practical assessment of cognitive status in geriatric patients. It is used as a brief screening tool for cognitive impairment and does not identify specific disorders. It concentrates only on the cognitive aspects of mental functions and excludes questions on mood, abnormal mental experiences as well as the form of thinking.
Beck depression inventory (BDI) | easily administered and requires only 5-10 minutes to complete depending on the impairment of the individual
  • The BDI-II contains 21 items on a 4-point scale from 0 (symptom absent) to 3 (severe symptoms). Anxiety symptoms are not assessed but affective, cognitive, somatic, and vegetative symptoms are covered, reflecting the DSM-IV criteria for major depression. Scoring is achieved by adding the highest ratings for all 21 items. The minimum score is 0 and maximum score is 63. Higher scores indicate greater symptom severity.
.Katz Index of Independence in Activities of Daily Living | easily administered and requires only 5-10 minutes to complete depending on the impairment of the individual
  Katz ADL is the most appropriate instrument to assess functional status as a measurement of the client's ability to perform activities of daily living independently. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding.

CONTACTS AND LOCATIONS:
Overall Officials: Hossam M Mohammed, PHD, Principal Investigator — Cairo University
Locations (1):
- Faculty of physical therapy .Cairo university, Cairo, Egypt